CLINICAL TRIAL: NCT00707330
Title: A Randomized, Single Blinded, Open-Label Crossover-Study of the Possible Induction of Oxidative Stress by Clarithromycin in Healthy Subjects
Brief Title: Study of the Ability of Clarithromycin to Induce Oxidative Stress
Acronym: CLAROX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Henrik Enghusen Poulsen, professor, dr. med., overlæge, Head of Department of Clinical Parmacology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 3-12-1-18-15-23; EudraCT 2008-001299-61; VEK H-D-2008-026; DKMA 2612-3720; Datatilsynet 2008-41-2030
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Oxidative Stress
Keywords: oxidative stress; 8-oxo-deoxyguanine; 8-oxodG; clarithromycin; malondialdehyde; mda; vitamine C; ascorbic acid
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects randomised to this arm will first be treated with Clarithromycin for a week, then have a 2-week washout, and finally one week of no treatment
  Interventions: Drug: Clarithromycin
- 2 (Active Comparator): Subjects randomised to this arm will first receive one week of no treatment, then have a 2-week washout, and finally be treated with Clarithromycin for a week
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — Prolonged release tablet, 500 mg, 1 tablet a day for a week
  Other Names: Klacid Uno; ATC: J01FA09

SUMMARY:
The purpose of the study is to examine whether Klacid® (Clarithromycin) will induce oxidative stress (stress from oxygen) in healthy subjects. This is done by measuring the content of a particular substance in the urine sample, which is released when the body is exposed to oxidative stress. In addition, there will also be taken blood samples, which is analysed for another substance that is indicative of oxidative stress.

DETAILED DESCRIPTION:
The purpose of the study is to examine whether Klacid® induce oxidative stress in healthy subjects.

Many studies have shown that atherosclerosis can cause acute myocardial infarction (AMI). The development of atherosclerosis is exacerbated by simultaneous infection with Chlamydophila pneumoniae, and its accompanying inflammation. There has been shown a positive association between Chlamydophila pneumoniae antibodies and the incidence of cardiovascular complications, suggesting that Chlamydophila pneumoniae could exacerbate the development of atherosclerosis [1]. It has therefore been tried to treat atherosclerotic AMI- patients prophylactically with macrolide antibiotics (which is used to treat Chlamydia infections), to halt development of the atherosclerosis and the accompanying risk of a new acute myocardial infarction.

Two minor studies have demonstrated a positive effect of macrolide-treatment, why a major Danish study of Clarithromycin was implemented [2-4]. Clarithromycin treatment was tested against placebo in 4373 atherosclerotic patients who had had an AMI. It appeared that the use of clarithromycin led to an increased cardiovascular mortality, which could not be explained [4]. The finding of the study suggests that clarithromycin cannot be used for secondary prophylaxis of cardiovascular complications, but whether clarithromycin can be used for primary prophylaxis is not known.

It has been shown that oxidative stress can participate in the development of cardiovascular complications [5], and it could be such an oxidative stress that had led to the increased mortality in the above study. Especially because a recent american study found evidence that bactericidal antibiotics induce oxidative stress in bacteria, leading to cell death [6]. This oxidative stress contributes significantly to the impact of the bactericidal antibiotics, which was thought to be primarily attributed to their specific drug/target interactions. The same study also examined erythromycin, from which clarithromycin is a derivate. Erythromycin showed no induction of oxidative stress, but clarithromycin is twice as effective as erythromycin, which could be due to oxidative stress caused by clarithromycin.

This study seeks to clarify a possible mechanism for clarithromycin, by an examination on healthy volunteers without atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Non-smoker
* Body mass index (BMI) must be ≥18 and ≤ 30
* Blood pressure must be within the following limits:
* Systolic blood pressure (110 mmHg > X < 140 mmHg)
* Diastolic blood pressure (60 mmHg > Y < 90 mmHg)
* Normal lipid plasma levels:
* Total cholesterol (≤ 6,0 mmol/l)
* HDL-cholesterol (≥ 0,9 mmol/l)
* LDL-cholesterol (≤ 4,5 mmol/l)
* Triglycerides (0,5-2,2 mmol/l)

Exclusion Criteria:

* Smokers
* CRP: > 10 mg/l
* Prolonged QT interval (defined as QTc > 450 msec.)
* Severe renal insufficiency (Cpl (creatinine) > 0100 mmol/l)
* Hereditary galactose intolerance
* A special form of hereditary lactase deficiency (Lapp Lactase deficiency)
* Glucose/galactose malabsorption
* Use of medicines and herbal remedies that affect/is affected by Clarithromycin, or lead to QT prolongation, for example, cisapride, pimozide, terfenadine, ergotamine, dihydroergotamine, fluconazole, ritonavir, carbamazepine, kinidin, disopyramide, lovastatin, simvastatin, warfarin, acenocoumarol, sildenafil, Tadalafil, vardenafil, theophylline, tolterodine, triazolo benzodiazepins, omeprazole, colchinine, digoxin, zidovudine, phenytoin, valproat, atazanavir, itraconazole, saquinavir
* Inborn condition with prolonged QT interval
* The following disorders:
* Coronary artery disease
* Former cardiac arrhythmias
* Severe heart insufficiency
* Non-compensated hypokalemia (defined as Cpl (K) < 3.2 mmol/ l) and/or hypomagnesemia (defined as Cpl (Mg) < 0.67 mmol/l)
* Bradycardia ( < 50 bpm)
* Known allergy to clarithromycin or other macrolides
* Narcotic
* Eating food supplements

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Amount of 8-oxo-deoxyguanine in 24 hour-urine measured in nmol/mmol creatinine | End of study (July-August 2008)
Amount of Malondialdehyde in plasma | End of study (July-August 2008)

SECONDARY OUTCOMES:
Amount of Total Vitamin C (Ascorbic acid) in plasma | End of study (July-August 2008)
Caffeine-metabolite ratio in 24 hour-urine | End of Study (July-August 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik E Poulsen, dr. med., Principal Investigator — Head of Department, Department of Clinical Pharmacology, Rigshospitalet
Locations (1):
- Department of Clinical Pharmacology Q, Rigshospitalet, Blegdamsvej 9, Kopenhagen O, Denmark

REFERENCES:
- [Background] Muhlestein JB, Anderson JL. Infectious serology and atherosclerosis: how burdensome is the risk? Circulation. 2003 Jan 21;107(2):220-2. doi: 10.1161/01.cir.0000043909.78380.a0. No abstract available. PMID 12538417
- [Background] Gupta S, Leatham EW, Carrington D, Mendall MA, Kaski JC, Camm AJ. Elevated Chlamydia pneumoniae antibodies, cardiovascular events, and azithromycin in male survivors of myocardial infarction. Circulation. 1997 Jul 15;96(2):404-7. doi: 10.1161/01.cir.96.2.404. PMID 9244203
- [Background] Gurfinkel E, Bozovich G, Daroca A, Beck E, Mautner B. Randomised trial of roxithromycin in non-Q-wave coronary syndromes: ROXIS Pilot Study. ROXIS Study Group. Lancet. 1997 Aug 9;350(9075):404-7. doi: 10.1016/s0140-6736(97)07201-2. PMID 9259655
- [Background] Jespersen CM, Als-Nielsen B, Damgaard M, Hansen JF, Hansen S, Helo OH, Hildebrandt P, Hilden J, Jensen GB, Kastrup J, Kolmos HJ, Kjoller E, Lind I, Nielsen H, Petersen L, Gluud C; CLARICOR Trial Group. Randomised placebo controlled multicentre trial to assess short term clarithromycin for patients with stable coronary heart disease: CLARICOR trial. BMJ. 2006 Jan 7;332(7532):22-7. doi: 10.1136/bmj.38666.653600.55. Epub 2005 Dec 8. PMID 16339220
- [Background] Dhalla NS, Temsah RM, Netticadan T. Role of oxidative stress in cardiovascular diseases. J Hypertens. 2000 Jun;18(6):655-73. doi: 10.1097/00004872-200018060-00002. PMID 10872549
- [Background] Kohanski MA, Dwyer DJ, Hayete B, Lawrence CA, Collins JJ. A common mechanism of cellular death induced by bactericidal antibiotics. Cell. 2007 Sep 7;130(5):797-810. doi: 10.1016/j.cell.2007.06.049. PMID 17803904